CLINICAL TRIAL: NCT00747253
Title: AutoLITT™ FIM Trial - A Prospective First-In-Man (FIM) Safety Trial of the AutoLITT Laser Treatment of Recurrent/Progressive Brain Tumors
Brief Title: Monteris AutoLITT™ FIM Safety Trial for Recurrent/Progressive Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Monteris Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AutoLITT™ FIM
Record Dates: First submitted 2008-09-02; First posted 2008-09-05 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Brain Tumor; Brain Tumor, Recurrent; Brain Neoplasm; Brain Cancer; Glioblastoma Multiforme; Recurrent Glioblastoma Multiforme
Keywords: laser interstitial thermal therapy; laser therapy; thermal therapy; brain tumors; recurrent brain tumor; progressive brain tumor; glioblastoma multiforme tumor
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Active Arm (Experimental): Only Arm. Patients treated using AutoLITT System.
  Interventions: Device: AutoLITT system

INTERVENTIONS:
Device: AutoLITT system — laser treatment with the AutoLITT system

SUMMARY:
The main purpose of this study is to evaluate the safety and performance of the AutoLITT system for the treatment of recurrent/progressive glioblastoma multiforme tumors (GBM).

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of GBM treated with radiotherapy with or without surgical resection and/or chemotherapy
* Clinical/radiographic suspicion of tumor recurrence/progression

Exclusion Criteria:

* Previous treatment of target GBM with stereotactic radiosurgery, brachytherapy, or carmustine impregnated wafers (Gliadel).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is safety, as determined by absence of severe clinical toxicity or procedure-related neurological deficits | 14 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gene Barnett, MD, Principal Investigator — The Cleveland Clinic; Andrew Sloan, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, 9500 Euclid Ave, Cleveland, Ohio

REFERENCES:
- [Derived] Sloan AE, Ahluwalia MS, Valerio-Pascua J, Manjila S, Torchia MG, Jones SE, Sunshine JL, Phillips M, Griswold MA, Clampitt M, Brewer C, Jochum J, McGraw MV, Diorio D, Ditz G, Barnett GH. Results of the NeuroBlate System first-in-humans Phase I clinical trial for recurrent glioblastoma: clinical article. J Neurosurg. 2013 Jun;118(6):1202-19. doi: 10.3171/2013.1.JNS1291. Epub 2013 Apr 5. PMID 23560574